CLINICAL TRIAL: NCT00785317
Title: Effects of Oral 1 mg Oestradiol (E2)/ 2 mg of Drospirenone (DRSP) Compared to Oral 1 mg of Oestradiol (E2)/ 0.5 mg Noresthisterone Acetate (NETA)on the Postmenopausal Breast; a Double Blind Randomized Prospective Study
Brief Title: Effects of Estradiol on Menopausal Breast
Acronym: BrAVA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Eva Lundström, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080818
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Hormone Replacement Therapy
Keywords: Postmenopausal Hormone Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angemin (Experimental): 1 mg of oral oestradiol (E2) in continuous combination with 2 mg of DRSP
  Interventions: Drug: Angemin vs Activelle
- Activelle (Active Comparator): 1 mg of oral E2 in continuous combination with 0.5 mg of NETA
  Interventions: Drug: Angemin vs Activelle

INTERVENTIONS:
Drug: Angemin vs Activelle — 1 mg of oral oestradiol (E2) in continuous combination with 2 mg of DRSP or 1 mg of oral E2 in continuous combination with 0.5 mg of NETA during six months.

SUMMARY:
The purpose of this study is to evaluate the effects on breast in postmenopausal women randomized to either oestradiol in combination with DRSP or E2 in combination with NETA during six months.

ELIGIBILITY:
Inclusion Criteria:

* Naturally postmenopausal, symptomatic, apparently healthy women, with the need for hormone therapy aged 50 - 70 years with a BMI >18 and ≤30 kg/m2 and without any previous history of breast disease will be recruited for the study.
* They should be amenorrheic for at least 12 months or less than 12 months with S- FSH values >40 IU/L.
* They should be free of any sex hormone treatment for at least three months before inclusion.

Exclusion Criteria:

* General contraindications for HT according to Swedish product label. Age >60 years. BMI ≤18 or ≥30 kg/m2.
* Any previous history of cancer.
* Any previous history of breast disease or abnormal mammogram.
* In addition: hypertension (systolic BP >160 mm Hg or diastolic >100 mm Hg), hyperlipidemia (total cholesterol >8.0 mmol/L or triglycerides >3.0 mmol/L), diabetes mellitus, history of thromboembolic disease, heart failure, liver disease or porphyria, undiagnosed vaginal bleeding. No sex hormone treatment for at least three months before inclusion.
* No concomitant treatment known to influence hormone metabolism (warfarin, rifampicin, carbamazepine, griseofulvin, hydantoins, primidone, barbiturates, broad spectrum antibiotics) is to be accepted.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-10 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Mammographic breast density - classified according to digitized data-based quantification of breast density. | 6 months

SECONDARY OUTCOMES:
Effects on serum levels of Oestradiol etc. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden